CLINICAL TRIAL: NCT04532593
Title: A Randomized, Placebo Controlled, Single-blinded Clinical Trial to Evaluate the Efficiency of Autologous Adipose Stem Cell in Promoting Skin Graft
Brief Title: Autologous Adipose Stem Cell Assisted Skin Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Huaxi Hospital (Other); Ruijin Hospital (Other); Shanghai Zhongshan Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Qing-FengLi Li,MD, Director, Professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH9H-2020-T185-1
Record Dates: First submitted 2020-08-21; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Skin Graft
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stem cell group (Experimental)
  Interventions: Procedure: autologous adipose stem cell injection
- Control (Placebo Comparator)
  Interventions: Procedure: saline injection

INTERVENTIONS:
Procedure: autologous adipose stem cell injection — Abdominal or buttock fat will be aspirated under local anesthesia or general anesthesia by conventional methods (0.5 ml fat was aspirated per 1 cm2 of skin graft area). The matrix component rich in adipose stem cells will be obtained by chopping, washing and centrifugation. The intervention treatment will be performed after the skin graft sutured. The stem cell components will be injected underneath the skin graft (0.05 ml/cm2).
  Arms: Stem cell group
Procedure: saline injection — saline will be injected underneath skin graft (0.05 ml/cm2).
  Arms: Control

SUMMARY:
Skin graft is a commonly used method in wound repair. The long-term outcome of skin graft is unsatisfied because of the complications of contraction, pigmentation and stiffness. In our preclinical researches, we found that adipose stem cell can improve the texture of grafted skin and reduce contraction. In this trial, we will evaluate the efficiency and safety of autologous adipose stem cells in improving skin graft outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 6-70 years old;
2. Gender: male and female;
3. Scar, surface tumor or soft tissue defect evaluated to be suitable for skin grafting;
4. With two skin grafting areas and the edges more than 4cm apart;
5. Sign informed consent, participate in the study and be able to cooperate with the follow-up.

Exclusion Criteria:

1. Those who are not suitable for skin grafting;
2. There who are with local lesions in the operation area, such as infection, blood supply disturbance, delayed healing history, decreased soft tissue vitality, history of radiotherapy or going to receive radiotherapy, active ulcer, etc;
3. With severe medical diseases (such as diabetes, hepatitis, coronary heart disease, arteriosclerosis, glomerulonephritis, autoimmune diseases, etc.) were complicated;
4. Those who are receiving anticoagulant therapy and cannot suspend treatment;
5. Those who are with abnormal blood routine test, abnormal coagulation function, abnormal cardiac function, abnormal liver function or renal function evaluated by researchers according to the laboratory examination and other clinical signs and symptoms,
6. Those who can't tolerate the operation risk according to the surgeon's evaluation;
7. Pregnant and lactating women;
8. Those who have mental illness, have no insight, can not express and cooperate with each other;
9. Participant in other clinical trials within 30 days before the screen visit of this trial;
10. Those who have not signed the informed consent.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Skin elasticity | 6 months
  Skin elasticity analyzed by Cutometer. The R2 value is used to evaluated the skin elasticity.

SECONDARY OUTCOMES:
Skin elasticity | 3 months
  Skin elasticity analyzed by Cutometer. The R2 value is used to evaluated the skin elasticity.
Skin elasticity | 12 months
  Skin elasticity analyzed by Cutometer. The R2 value is used to evaluated the skin elasticity.
Skin color | 3 months
  Skin color analyzed by CK Colorimeter CL400. The iTA value is used to evaluate the color of skin graft.
Skin color | 6 months
  Skin color analyzed by CK Colorimeter CL400. The iTA value is used to evaluate the color of skin graft.
Skin color | 12 months
  Skin color analyzed by CK Colorimeter CL400. The iTA value is used to evaluate the color of skin graft.
POSAS questionnaire of patient | 3 months
  POSAS questionnaire of patient. Five questions of pain, itch, thickness, color, stiffness, irregularity. Each question ranks 0, 1, 2. Total score is 0 to 10.
POSAS questionnaire of patient | 6 months
  POSAS questionnaire of patient. Five questions of pain, itch, thickness, color, stiffness, irregularity. Each question ranks 0, 1, 2. Total score is 0 to 10.
POSAS questionnaire of patient | 12 months
  POSAS questionnaire of patient. Five questions of pain, itch, thickness, color, stiffness, irregularity. Each question ranks 0, 1, 2. Total score is 0 to 10.
POSAS questionnaire of investigator | 3 months
  POSAS questionnaire of investigator. Six questions of vascularity, pigmentation, texture, thickness, pliability, surface area. Each question ranks 0, 1, 2. Total score is 0 to 12.
POSAS questionnaire of investigator | 6 months
  POSAS questionnaire of investigator. Six questions of vascularity, pigmentation, texture, thickness, pliability, surface area. Each question ranks 0, 1, 2. Total score is 0 to 12.
POSAS questionnaire of investigator | 12 months
  POSAS questionnaire of investigator. Six questions of vascularity, pigmentation, texture, thickness, pliability, surface area. Each question ranks 0, 1, 2. Total score is 0 to 12.